CLINICAL TRIAL: NCT06911749
Title: Contrast Enhanced Multispectral Optoacoustic Tomography and MRI for Non-invasive Assessment of Intestinal Transit Time in Children With Chronic Bowel Emptying Disorders
Brief Title: MSOT and MRI for Non-invasive Assessment of Intestinal Transit Time in Children With Chronic Bowel Emptying Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. med. Sonja Diez (Other)
Responsible Party: Sponsor-Investigator, Dr. med. Sonja Diez, PD Dr. med. Sonja Diez, Friedrich-Alexander-Universität Erlangen-Nürnberg
Organization: Friedrich-Alexander-Universität Erlangen-Nürnberg (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 24-373-B; Ethics Committee FAU (Other: Universitätsklinikum Erlangen (Friedrich-Alexander Universität))
Record Dates: First submitted 2025-02-25; First posted 2025-04-04 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-03

CONDITIONS: Chronic Constipation; Slow Transit Constipation; Intestinal Transit Disorder; Hirschsprungs Disease
Keywords: slow transit constipation; MSOT; ICG; gastrointestinal transit; Hirschsprungs Disease
MeSH Terms: conditions — Hirschsprung Disease

STUDY DESIGN:
Intervention Model Description: This study is a monocentric observational study with prospective data collection. It is conducted as an Investigator-Initiated Trial (IIT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Active Comparator): The control group consists of young, healthy adults without bowel emptying disorders. The aim of this group is to provide baseline measurements for gastrointestinal transit time and peristalsis using Multispectral Optoacoustic Tomography (MSOT) and MRI, allowing for comparison with the intervention group and ensuring the reliability of the diagnostic approach.
  Interventions: Diagnostic Test: MSOT with ICG; Diagnostic Test: MRI
- Transit Disorder Group (Active Comparator): The intervention group consists of pediatric patients suffering from chronic defecation disorders, including idiopathic chronic constipation, slow transit constipation (STC), and outlet obstruction (OO). The aim of the intervention is to assess gastrointestinal transit time and peristalsis using a novel, non-invasive combination of Multispectral Optoacoustic Tomography (MSOT) and MRI.
  Interventions: Diagnostic Test: MSOT with ICG; Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MSOT with ICG — Application of Multispectral Optoacoustic Tomography (MSOT) in combination with the oral contrast agent Indocyanine Green (ICG) to measure gastrointestinal transit time
Diagnostic Test: MRI — Non-invasive MRI imaging technique will be employed to assess the peristalsis of intestinal segments

SUMMARY:
The project presented here is a monocentric clinical study conducted by the Pediatric Surgery and Pediatrics departments of the University Hospital Erlangen. The study aims to experimentally expand the diagnostic approach for patients aged 0-17 years suffering from chronic bowel emptying disorders, regardless of any underlying causal or previously treated conditions.

At the core of this clinical study is the application of Multispectral Optoacoustic Tomography (MSOT) in combination with the oral contrast agent Indocyanine Green (ICG) to measure gastrointestinal transit time in children. Unlike conventional X-ray diagnostics, MSOT is radiation-free and considered non-invasive, although it has not yet been standardized for routine clinical use. Additionally, a contrast-free, non-invasive MRI technique will be employed to assess the peristalsis of intestinal segments.

The study aims to standardize the collection and evaluation of patient data following the administration of ICG and subsequent measurements using MSOT and MRI. The objective is to assess gastrointestinal transit time and peristalsis and, ultimately, to optimize therapy for affected patients. This is of particular importance in the coloproctology specialist consultation within the Pediatric Surgery and Pediatrics departments, as follows:

It enables differentiation between patients with slow transit constipation and outlet obstruction.

It allows for a more targeted application and evaluation of neuromodulation therapy, which is used within clinical studies.

This approach allows for the identification of specific intestinal segments with delayed transit time, enabling targeted electrical stimulation of these regions.

A control group of healthy adult volunteers will participate in the study on a voluntary basis.

DETAILED DESCRIPTION:
The term chronic defecation disorders encompasses a wide range of conditions in the current medical literature. Among them, idiopathic chronic constipation represents the central subgroup of patients, often suffering from therapy-refractory symptoms. However, other causes of chronic defecation disorders must also be considered, such as Hirschsprung's disease, cystic fibrosis, congenital malformations and their postoperative complications, or neurogenic bladder and rectal emptying disorders. Additionally, chronic fissures, congenital anal stenosis, and previous abdominal surgeries can contribute to chronic defecation disorders.

In most cases, the underlying cause is not a single, well-controlled symptom but rather a heterogeneous symptom complex. Chronic constipation, for instance, is defined based on various symptoms as per the Rome IV criteria, requiring a duration of at least three months for diagnosis. In children, this condition frequently presents as a combination of defecation difficulties, severe abdominal pain, food refusal, encopresis, enuresis, and reduced activity levels, often necessitating a multimodal and sometimes highly burdensome therapy. Patients typically experience significant distress and markedly reduced quality of life.

The prevalence of chronic constipation in children and adolescents is high, with reported rates reaching up to 34%. However, in more than 90% of cases, no organic cause can be identified. Conservative treatment approaches are often inadequate or fail to prevent long-term chronicity. Despite this, defecation disorders in children and adolescents are frequently underestimated and sometimes managed within psychiatric treatment settings, which may lead to long-term physical and psychological developmental impairments.

Diagnostic Challenges

Following the exclusion of manifest organic causes, the differentiation between "slow transit constipation" (STC) and "outlet obstruction" (OO) remains a major diagnostic challenge in children. Further complicating matters, many pediatric patients exhibit mixed forms of both conditions.

Slow transit constipation (STC) is characterized by a generalized delay in bowel transit, with predominantly genetic but also other organic causes. This condition arises from innervation disorders of the intestine, dysfunctions of the autonomic nervous system, abnormalities in the smooth muscle layers of the intestinal wall, as well as endocrine and metabolic dysfunctions. Typical symptoms include severe constipation, chronic abdominal pain, and therapy-resistant fecal incontinence.

Outlet obstruction (OO), in contrast, is caused by impaired stool evacuation at the anal level, often due to dyssynergic defecation or, less commonly, anatomical obstructions. Currently, a definitive differentiation between STC and OO in clinical practice is rarely performed, as non-invasive diagnostic tools are lacking. The only gold-standard diagnostic procedure available is anorectal manometry, which requires patient cooperation, making it impractical for young children. Additionally, the rectal insertion of probes and balloons renders it an invasive and potentially traumatizing procedure, which can exacerbate symptoms. As a result, a minimum patient age is required, and the findings are often difficult to interpret objectively.

Existing Methods for Transit Time Measurement

The delayed intestinal transit time associated with STC can be evaluated using:

The modified Hinton test Motility capsules Gastrointestinal transit scintigraphy The lactulose hydrogen breath test

In Germany, the modified Hinton test remains the gold standard. This involves ingestion of 10 radiopaque markers per day for six consecutive days, followed by an abdominal X-ray on day seven to calculate the oro-anal transit time. However, this method is time-consuming and should be used with caution in children due to radiation exposure. Other emerging methods include:

SmartPill motility capsules, which measure temperature, pH, and intraluminal pressure to determine total transit time. However, these are not commercially available and do not offer significant advantages over conventional transit studies to justify the additional cost.

Gastrointestinal transit scintigraphy, which involves a technetium-labeled meal and subsequent gamma camera imaging at 1, 2, and 4 hours. However, this method is time-intensive, expensive, and not widely available. Additionally, it is considered invasive and unsuitable for pediatric use due to radiation exposure.

The lactulose hydrogen breath test, which measures the oro-cecal transit time by detecting bacterial fermentation of lactulose in the cecum. However, this method is limited to assessing small bowel transit only.

Notably, none of these tests can differentiate between an organic and a functional cause of constipation.

Multispectral Optoacoustic Tomography (MSOT) for Transit Time Measurement

Multispectral optoacoustic tomography (MSOT) is based on the emission of laser light at multiple near-infrared wavelengths. This light stimulates biological tissue, leading to ultrasound wave emission, which is then reconstructed into an image. MSOT enables the acquisition of both single-wavelength images and spectrally unmixed images, allowing for the visualization of molecules with known absorption properties, such as hemoglobin and lipids.

Contrast-enhanced MSOT (CE-MSOT) allows for non-invasive, radiation-free visualization of chyme passage through the gastrointestinal tract. Studies have demonstrated that orally administered Indocyanine Green (ICG) can be detected at various locations within the GI tract-including the gastric antrum, terminal ileum, and sigmoid colon-using MSOT.

ICG, which has an absorption peak at approximately 800 nm in the near-infrared spectrum, is well-suited for optical imaging techniques. It is already widely used in medical applications, including intraoperative imaging, liver function diagnostics, and cardiovascular assessments.

Although the oral administration of ICG is an off-label use, systemic side effects are highly unlikely, as ICG is not absorbed and does not undergo enterohepatic circulation, according to its official drug information.

The complete gastrointestinal passage of ICG has been confirmed through fluorescence microscopy detection of ICG in stool samples from subjects following oral administration. Based on this methodology, this study aims to evaluate intestinal transit time in patients with chronic defecation disorders, providing a novel, non-invasive diagnostic tool to address the current gap in pediatric gastrointestinal transit assessment.

Study Objective: Combining MSOT and MRI for Comprehensive GI Transit Analysis

This study aims to integrate MRI sequences specifically designed to visualize peristaltic bowel movements with high temporal resolution, allowing for a detailed assessment of peristaltic frequency and patterns across different intestinal segments. By capturing these peristaltic movements, it becomes possible to identify abnormally reduced peristalsis in the pediatric patient cohort.

By combining MSOT-derived transit time measurements with MRI-based peristalsis visualization, this study offers a comprehensive and non-invasive method to assess gastrointestinal motility. Through this approach, it will be possible to detect segments of the intestine with abnormal transit times and assess chyme transport throughout the entire gastrointestinal tract without exposing patients to radiation or invasive procedures.

ELIGIBILITY:
Inclusion Criteria:

Patient Group

* Written informed consent from the participant (starting at age 6).
* Written informed consent from the legal guardian(s).
* Suspected or confirmed diagnosis of chronic defecation disorder.
* Age ≤ 18 years.
* Willingness and ability to participate, with sufficient German language skills to understand the informed consent document.

Control Group

* Written informed consent from the participant.
* Age > 18 years.
* BMI < 25 or medical suitability for MSOT examination as assessed by a physician.
* Willingness and ability to participate, with sufficient German language skills to understand the informed consent document.

Exclusion Criteria:

* Age < 1 year.
* Pregnancy or breastfeeding.
* Tattoos in the examination area.
* Subcutaneous fat tissue thickness > 3 cm.
* Known hypersensitivity to ICG, sodium iodide, or iodine.
* Thyroid dysfunction, including hyperthyroidism or focal/diffuse thyroid autonomy.
* Recent thyroid function testing with radioactive iodine treatment (within two weeks before or after the study).
* Impaired renal function.
* Use of specific medications, including:

  * Beta-blockers,
  * Anticonvulsants,
  * Cyclopropane,
  * Bisulfite compounds,
  * Haloperidol,
  * Heroin,
  * Meperidine,
  * Metamizole,
  * Methadone,
  * Morphine,
  * Nitrofurantoin,
  * Opium alkaloids,
  * Phenobarbital,
  * Phenylbutazone,
  * Probenecid,
  * Rifamycin,
  * Any injection containing sodium bisulfite.
* General contraindications for MRI, such as electrical implants (e.g., pacemakers, perfusion pumps).
* Severe claustrophobia preventing MRI examination.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
ICG signal intensitiy | From enrollment to the end of measurements after one week
  Measurement of qualitative and quantitative ICG signal within the lumen of the GI tract, expressed in arbitrary units (AU).
MRI-Based Diagnostic Image Quality | From enrollment to the end of measurements after one week
  Assessment of overall MRI image quality using a standardized grading scale.
MRI Motion Robustness | Time Frame: From enrollment to the end of measurements after one week.
  Evaluation of motion artifacts in MRI imaging, scored on a predefined motion robustness scale.
MRI-Based Peristalsis Frequency | Time Frame: From enrollment to the end of measurements after one week
  Measurement of peristaltic contractions per minute in different intestinal segments.
MRI-Based Peristalsis Amplitude | Time Frame: From enrollment to the end of measurements after one week.
  Quantification of bowel wall movement amplitude in millimeters (mm).

SECONDARY OUTCOMES:
Single-Wavelength Optoacoustic Signal | From enrollment to the end of measurements after one week
  Quantitative assessment of single-wavelength optoacoustic measurements, expressed in arbitrary units (AU).
Optoacoustic Spectrum Analysis | From enrollment to the end of measurements after one week
  Comprehensive optoacoustic signal analysis across multiple wavelengths, normalized in arbitrary units (AU).
Ultrasound imaging | From enrollment to the end of measurements after one week
  Ultrasound imaging with assement of the presence of stool.
Gastrointestinal Symptom Assessment | From enrollment to the end of the study after one year.
  Evaluation of symptom severity, including abdominal pain, nausea, diarrhea, and other gastrointestinal complaints, recorded on a standardized symptom severity scale.
Demographic parameters | From enrollment to the end of measurements after one week
  Collection of demographic data, including age (years), height (cm), weight (kg), and other relevant characteristics.

OTHER OUTCOMES:
Blood Test Results and Medical Findings | From enrollment to the end of the study after one year
  Analysis of laboratory test results and clinical findings extracted from medical records.
Pediatric Surgery Database Analysis | From enrollment to the end of the study after one year.
  Processing and evaluation of patient data from the specialized outpatient clinic for chronic defecation disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Diez, PD Dr. med., Principal Investigator — Friedrich-Alexander-Universität Erlangen-Nürnberg; Adrian Regensburger, PD Dr. med., Principal Investigator — Friedrich-Alexander-Universität Erlangen-Nürnberg
Locations (1):
- University Hospital Erlangen, Pediatric Surgery, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paulus LP, Buehler A, Wagner AL, Raming R, Jungert J, Simon D, Tascilar K, Schnell A, Rother U, Eckstein M, Lang W, Hoerning A, Schett G, Neurath MF, Waldner MJ, Trollmann R, Woelfle J, Bohndiek SE, Regensburger AP, Knieling F. Contrast-Enhanced Multispectral Optoacoustic Tomography for Functional Assessment of the Gastrointestinal Tract. Adv Sci (Weinh). 2023 Aug;10(23):e2302562. doi: 10.1002/advs.202302562. Epub 2023 Jun 8. PMID 37289088